CLINICAL TRIAL: NCT00793871
Title: A Single-arm, Open-label, Multi-center, Phase Iv, Efficacy And Safety Study Of Sunitinib Malate In The Treatment Of Chinese Patients With Gastrointestinal Stromal Tumor After Disease Progression On Or Intolerance To Imatinib Mesylate
Brief Title: Safety And Efficacy Study Of Sunitinib Malate In Chinese Patients With Imatinib Resistant Or Intolerant Malignant Gastrointestinal Stromal Tumor
Acronym: GIST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181177
Record Dates: First submitted 2008-11-17; First posted 2008-11-19 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-10

CONDITIONS: Gastrointestinal Neoplasms, Gastrointestinal Stromal Tumors
Keywords: sunitinib; Phase IV; gastrointestinal stomal tumor; imatinib resistant or intolerant; Chinese
MeSH Terms: conditions — Gastrointestinal Neoplasms; Gastrointestinal Stromal Tumors | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sunitinib (Experimental): single agent sunitinib, single arm
  Interventions: Drug: Sunitinib Malate (SU011248)

INTERVENTIONS:
Drug: Sunitinib Malate (SU011248) — Subjects will receive treatment with sunitinib in repeated 6-week cycles (4 weeks on, 2 weeks off), at a starting dose of 50 mg.

SUMMARY:
To investigate safety and efficacy of single agent sunitinib malate in Chinese Patients With Imatinib Resistant Or Intolerant Malignant Gastrointestinal Stromal Tumor.

ELIGIBILITY:
Inclusion Criteria:

* Histologically-proven diagnosis of malignant GIST (Gastrointestinal Stromal Tumors).
* Evidence of unidimensionally measurable disease
* Failure of prior treatment with imatinib or intolerant to imatinib
* Male or female, 18 years of age or older.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.
* Resolution of all acute toxic effects
* Adequate organ function.

Exclusion Criteria:

* Anticancer treatment after last dose of imatinib
* Major surgery within 4 weeks or radiation therapy within 2 weeks.
* Grade 3 hemorrhage within 4 weeks prior to starting the study treatment.
* Diagnosis of second malignancy within the last 5 years.
* History of brain disease.
* Cardiac disease within 12 months.
* Thyroid function abnormality.
* Ongoing cardiac dysrhythmias.
* Uncontrolled hypertension.
* Ongoing treatment with anticoagulant and CYP3A4 inhibitors and inducers.
* HIV or AIDS related illness.
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2014-04 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- China (4):
  - Nanjing Bayi Hospital, Nanjing, Jiangsu
  - Cancer Institute & Hospital Chinese Academy of Medical Sciences and PUMC, Beijing
  - Beijing Cancer Hospital, Beijing
  - 307 Hospital of PLA, Beijing

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181177

RESULTS

PARTICIPANT FLOW:
Groups:
- Sutent (Sunitinib Malate): The starting dose of sunitinib was 50 milligram (mg) orally once daily as a single agent for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks (schedule 4/2). Participants experiencing dose-limiting toxicity attributed to study medication had dose interrupted or reduced depending on individual tolerability. If dose reductions were required, the dose of 37.5 mg was achieved by administration of 3 × 12.5 mg capsules, and the dose of 25 mg was achieved by administration of 2 × 12.5 mg capsules. There was no limit for number of cycles for this study, study treatment was permanently discontinued upon disease progression, occurrence of unacceptable toxicity, withdrawal of participant consent, or another withdrawal criterion was met.
Period: Overall Study
Arm/Group | Sutent (Sunitinib Malate)
Started | 60
Received Treatment | 59
Completed | 0
Not Completed | 60
Not completed — Death | 50
Not completed — Lost to Follow-up | 3
Not completed — Study terminated by the Sponsor | 7

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who started study treatment.
Groups:
- Sutent (Sunitinib Malate): The starting dose of sunitinib was 50 mg orally once daily as a single agent for 4 consecutive weeks followed by a 2-week off-treatment period to form a complete cycle of 6 weeks (schedule 4/2). Participants experiencing dose-limiting toxicity attributed to study medication had dose interrupted or reduced depending on individual tolerability. If dose reductions were required, the dose of 37.5 mg was achieved by administration of 3 × 12.5 mg capsules, and the dose of 25 mg was achieved by administration of 2 × 12.5 mg capsules. There was no limit for number of cycles for this study, study treatment was permanently discontinued upon disease progression, occurrence of unacceptable toxicity, withdrawal of participant consent, or another withdrawal criterion was met.
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.1 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 39

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time (in weeks) from the date of the first treatment to the date of the first documentation of objective tumor progression or death due to any cause, whichever occurred first. Participants last known to be 1) alive, 2) on study treatment or discontinued study treatment, but haven't yet started a new anticancer treatment and 3) progression-free were censored at the date of the last objective disease assessment that verified lack of disease progression. Disease progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST version 1.0), as a >=20% increase in the sum of the longest dimensions of the target lesions taking as a reference the smallest sum of the longest dimensions recorded since the treatment started, or the appearance of one or more new lesions.
Time Frame: Baseline (Day 1) up to disease progression or death whichever occurred first (up to 264 weeks)
Population: Safety analysis included all participants who started study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
weeks | 46.4 [33.6 to 53.1]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (in weeks) from the date of the first treatment to the date of death due to any cause.
  In the absence of confirmation of death, survival time was censored at the last date the participant was known to be alive.
Time Frame: Baseline (Day 1) to death (up to 282 weeks)
Population: Safety analysis set included all participants who started study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
weeks | 111.3 [75.4 to 167.1]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the proportion of participants who achieved an objective response. A participant was considered to have an objective response if a confirmed best response of complete response (CR) or partial response (PR) was achieved according to RECIST, version 1.0. CR is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 millimeters (mm). PR is at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Baseline (Day 1) up to end of study treatment (up to 276 weeks)
Population: The per-protocol analysis set included all enrolled participants who had the disease under study, measurable disease and an adequate baseline disease assessment, and who started study treatment.
Measure: Number (95% Confidence Interval); unit: % of participants
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 58
% of participants | 19.0 [9.9 to 31.4]

4. Secondary Outcome: Time to Tumor Progression (TTP)
Description: TTP was defined as the time (in weeks) from the date of the first treatment to the date of the first documentation of objective tumor progression or death due to tumor progression. Participants last known to be 1) alive,2) on treatment or within 28 days of discontinuation from treatment and 3) progression-free were censored at the date of last objective disease assessment that verified lack of disease progression. Participants with no post baseline assessments were censored at the start date. Participants who died without prior objective disease progression and participants who discontinued treatment without objective disease progression within 28 days of last dose were censored at the date of the last objective disease assessment that verified lack of disease progression. Disease progression is defined using RECIST version 1.0.
Time Frame: Baseline (Day 1) up to objective tumor progression or death due to tumor progression (up to 264 weeks)
Population: Safety analysis set included all participants who started study treatment.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
weeks | 47.3 [34.1 to 59.3]

5. Other Pre Specified Outcome: Time to Tumor Response (TTR)
Description: TTR was defined as the time (in weeks) from the date of the first dose of study treatment to the date of the first documentation of objective tumor response (CR or PR based on RECIST, version 1.0) that was subsequently confirmed.
Time Frame: Baseline (Day 1) to tumor response (up to 82 weeks)
Population: All participants who started study treatment (safety analysis set) had a confirmed objective tumor response.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 11
weeks | 22.6 [10.4 to 57.3]

6. Secondary Outcome: Number of Participants With Abnormal Clinical Laboratory Measurements
Description: The total number of participants with laboratory test abnormalities without regard to baseline abnormality was assessed. Laboratory parameters included hematology (hemoglobin, platelets, white blood cell count, lymphocytes, neutrophils, basophils, eosinophils and monocytes), liver function (total bilirubin, aspartate aminotransferase, alanine aminotransferase, alkaline phosphatase, total protein and albumin), renal function (blood urea nitrogen, creatinine and uric acid), electrolytes (sodium, potassium, chloride, calcium, magnesium and phosphate), hormones (thyroxine and thyroid stimulating hormone), clinical chemistry (glucose), and urinalysis (urine protein) tests.
Time Frame: Baseline up to 28 days post last administration of study drug
Population: Safety analysis set included all participants who started study treatment.
Measure: Number; unit: participants
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
participants | 57

7. Secondary Outcome: Number of Participants With Significant Changes From Baseline in Physical Examination.
Description: Physical examinations including, but not limited to, general appearance, skin, neck, eyes, ears, nose, mouth, throat, breast, lungs, heart, abdomen, rectal, lymph nodes, extremities, thyroid, musculoskeletal, and nervous system were performed.
Time Frame: Baseline up to 28 days post last administration of study drug
Population: Safety analysis set included all participants who started study treatment.
Measure: Number; unit: participants
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
participants | 28

8. Secondary Outcome: Number of Participants With Significant Vital Signs Changes From Baseline
Description: Vital signs included blood pressure (BP), temperature, heart rate, respiration rate and body weight. The criteria for significant changes included BP: systolic BP (SBP) greater than (>) 150 millimeters of mercury (mm Hg) and/or diastolic BP (DBP) > 100 mm Hg, or SBP > 200 mm Hg and/or DBP > 110 mm Hg; temperature: >38.3 degrees Celsius (degrees C), or increase of greater than or equal to (>=)1.1 degrees C (baseline >=36.8 degrees C); heart rate: >120 beats per minute (bpm) or less than (<) 50 bpm, or increase of >=30 bpm or decrease of ≥30 bpm; respiration rate: > 40 /minute or < 8 /minute; weight: a change of 5% or more from baseline.
Time Frame: Baseline (Day 1) up to 28 days post last administration of study drug
Population: Safety analysis set included all participants who started study treatment.
Measure: Number; unit: participants
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
participants
  SBP >150 mm Hg or DBP >100 mm Hg | 9
  SBP >200 mm Hg or DBP >110 mm Hg | 1
  heart rate: <50 bpm | 0
  heart rate: >120 bpm | 0
  heart rate: >=30 bpm increase from baseline | 2
  heart rate: >=30 bpm decrease from baseline | 2
  temperature: >38.3°C | 0
  temperature: >=1.1°C increase (baseline >=36.8°C) | 0
  respiration rate: <8/minute | 0
  respiration rate: >40/minute | 0
  weight: >=5% increase from baseline | 12
  weight: >=5% decrease from baseline | 20

9. Secondary Outcome: Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG was used to assess participants' performance status: 0 (Fully active, able to carry on all pre-disease activities without restriction); 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work or office work); 2 (Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours); 3 (Capable of only limited self-care, confined to bed or chair more than 50% of waking hours); 4 (Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair); and 5 (Dead).
Time Frame: Baseline (Day 1), Last-on treatment visit (up to 28 days post last administration of study drug)
Population: Safety analysis set included all participants who started study treatment.
Measure: Number; unit: participants
Arm/Group | Sutent (Sunitinib Malate)
Number analyzed (Participants) | 59
participants
  Baseline, ECOG = 0 | 11
  Baseline, ECOG = 1 | 48
  Baseline, ECOG = 2 | 0
  Baseline, ECOG = 3 | 0
  Baseline, ECOG = 4 | 0
  Baseline, ECOG = 5 | 0
  Last on treatment, ECOG = 0 | 3
  Last on treatment, ECOG = 1 | 47
  Last on treatment, ECOG = 2 | 8
  Last on treatment, ECOG = 3 | 1
  Last on treatment, ECOG = 4 | 0
  Last on treatment, ECOG = 5 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Sutent (Sunitinib Malate)
Serious Adverse Events (participants affected / at risk) | 12/59
Other Adverse Events (participants affected / at risk) | 57/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sutent (Sunitinib Malate) (N=59)
Neutropenia (Blood and lymphatic system disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 3
Bile duct stenosis (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 1
Neuropathy peripheral (Nervous system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sutent (Sunitinib Malate) (N=59)
Anaemia (Blood and lymphatic system disorders) | 15
Leukopenia (Blood and lymphatic system disorders) | 38
Neutropenia (Blood and lymphatic system disorders) | 29
Thrombocytopenia (Blood and lymphatic system disorders) | 15
Hypothyroidism (Endocrine disorders) | 8
Eyelid oedema (Eye disorders) | 10
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 18
Mouth ulceration (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 8
Stomatitis (Gastrointestinal disorders) | 8
Vomiting (Gastrointestinal disorders) | 8
Face oedema (General disorders) | 3
Fatigue (General disorders) | 31
Pyrexia (General disorders) | 6
Hepatic function abnormal (Hepatobiliary disorders) | 3
Hyperbilirubinaemia (Hepatobiliary disorders) | 3
Nasopharyngitis (Infections and infestations) | 4
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 3
Alanine aminotransferase increased (Investigations) | 14
Aspartate aminotransferase increased (Investigations) | 21
Bilirubin conjugated increased (Investigations) | 3
Blood albumin decreased (Investigations) | 7
Blood alkaline phosphatase increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 13
Blood calcium decreased (Investigations) | 5
Blood chloride decreased (Investigations) | 4
Blood creatinine increased (Investigations) | 10
Blood glucose increased (Investigations) | 9
Blood lactate dehydrogenase increased (Investigations) | 5
Blood magnesium decreased (Investigations) | 5
Blood potassium decreased (Investigations) | 8
Blood urea increased (Investigations) | 13
Blood uric acid increased (Investigations) | 7
Gamma-glutamyltransferase increased (Investigations) | 3
Haemoglobin decreased (Investigations) | 23
Neutrophil count decreased (Investigations) | 22
Neutrophil percentage decreased (Investigations) | 9
Platelet count decreased (Investigations) | 26
Protein total decreased (Investigations) | 3
Protein urine present (Investigations) | 5
Weight decreased (Investigations) | 10
Weight increased (Investigations) | 3
White blood cell count decreased (Investigations) | 19
Decreased appetite (Metabolism and nutrition disorders) | 9
Hyperuricaemia (Metabolism and nutrition disorders) | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 9
Hypokalaemia (Metabolism and nutrition disorders) | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 8
Hyponatraemia (Metabolism and nutrition disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 3
Haematuria (Renal and urinary disorders) | 3
Proteinuria (Renal and urinary disorders) | 16
Hair colour changes (Skin and subcutaneous tissue disorders) | 7
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 30
Rash (Skin and subcutaneous tissue disorders) | 6
Skin discolouration (Skin and subcutaneous tissue disorders) | 20
Yellow skin (Skin and subcutaneous tissue disorders) | 5
Hypertension (Vascular disorders) | 17
Angina pectoris (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 1
Myocardial ischaemia (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 1
Sinus arrhythmia (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Conjunctival haemorrhage (Eye disorders) | 1
Dry eye (Eye disorders) | 1
Eyelash hyperpigmentation (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1
Chest discomfort (General disorders) | 1
Generalised oedema (General disorders) | 1
Hernia (General disorders) | 1
Mucous membrane disorder (General disorders) | 1
Oedema (General disorders) | 2
Oedema peripheral (General disorders) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Hepatic mass (Hepatobiliary disorders) | 1
Hepatomegaly (Hepatobiliary disorders) | 1
Jaundice (Hepatobiliary disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Lung infection (Infections and infestations) | 1
Pericoronitis (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood glucose decreased (Investigations) | 2
Blood sodium decreased (Investigations) | 1
Blood thyroid stimulating hormone increased (Investigations) | 2
Blood urine present (Investigations) | 2
C-reactive protein increased (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Glucose urine present (Investigations) | 1
Lymphocyte count decreased (Investigations) | 2
Platelet count increased (Investigations) | 1
Protein urine (Investigations) | 1
Red blood cell count decreased (Investigations) | 2
Red blood cells urine positive (Investigations) | 1
Thyroxine free decreased (Investigations) | 1
Thyroxine increased (Investigations) | 1
Tri-iodothyronine free decreased (Investigations) | 1
White blood cell count increased (Investigations) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Abdominal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebral haemorrhage (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Eating disorder (Psychiatric disorders) | 1
Haemoglobinuria (Renal and urinary disorders) | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 1
Nephritis (Renal and urinary disorders) | 2
Renal impairment (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Eczema (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.